CLINICAL TRIAL: NCT05552079
Title: Gaps In Awareness of Peripheral Arterial Disease in Hong Kong: A Cross Sectional Study
Brief Title: PAD Awareness Study
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Bryan Ping Yen YAN, Professor, Chinese University of Hong Kong
Other Study IDs: 2019.571
Record Dates: First submitted 2021-03-23; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Patients will be asked to show their consultation slip to confirm they attend to clinic on the day. The will also be asked to show their HKID card to comfirm they are aged 40 or above. The purpose of the study will be explained. If patient agrees to proceed, he/she will be given a self-administered questionniare. An interviewer-administered questionnaire will be provided for subjects who have poor sightedness or are illiterate. Since only anonymous data and no identifiable information will be collected, participants cannot be identified from the questionnaire. Therefore, inform consent will not be obtained.

SUMMARY:
Peripheral arterial disease (PAD) is one of the most common cardiovascular diseases in developed countries [1] and is an emerging problem in developing countries [2, 3]. The prevalence of PAD in European population studies ranged from 3.6 to 9.2 % and 10-20 % in those aged over 70 years [4]. In a recent meta-analysis, the prevalence of PAD in China increased gradually by age until mid-60s, after which the increase accelerated. In the early stages, PAD is mostly silent. With the progression of disease, it may manifest as intermittent claudication, pain at rest, non-healing ulcer and gangrene resulting in lower-extremity amputation [5]. PAD is a major cause of disability, loss of employment, and lifestyle changes, and is a marker for systemic atherosclerotic diseases. Patients with symptomatic PAD have at least a 30% risk of death within 5 years rising to almost 50% within 10 years, resulting primarily from myocardial infarction or stroke [4]. Despite the major health risks associated with PAD, it is generally not recognized by clinicians or the general public in comparison with other cardiovascular diseases. However, asymptomatic individuals also have higher risk of adverse cardiovascular events similar to those with symptomatic PAD [6]. Many studies have shown that public awareness of PAD is much lower than that of other diseases. It has been reported that awareness of PAD ranged from 20 to 36 %, whereas awareness of other common diseases was more than 60 % in the same population [6-9]. Awareness is important for patients and physicians, and the need for public awareness programs has been highlighted [10, 11]. There is paucity of published literature on public awareness of PAD in Asian countries. It is difficult to reduce the morbidity and mortality of untreated PAD without adequate public awareness of PAD and its risk factors and consequences [7]. Insights into public awareness of PAD will help in developing strategies for behavioral change communication and health promotion. In this study we aimed to assess awareness of PAD among adults in Hong Kong. The survey is designed to measure knowledge of factors that increase the risk for PAD and the clinical risk consequences of having PAD. These data will provide useful information to guide future local public cardiovascular educational efforts.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is one of the most common cardiovascular diseases in developed countries [1] and is an emerging problem in developing countries [2, 3]. The prevalence of PAD in European population studies ranged from 3.6 to 9.2 % and 10-20 % in those aged over 70 years [4]. In a recent meta-analysis, the prevalence of PAD in China increased gradually by age until mid-60s, after which the increase accelerated. In males, the prevalence of PAD ranged from 2.81% (95% CI = 1.77-4.43) in those aged 25-29 years to 21.95% (95% CI = 15.39-30.31) in those 95-99 years old. In females, the PAD prevalence increased from 3.84% (95% CI = 2.44-5.98) in those aged 25-29 years to 27.95% (95% CI = 20.14-37.37) in those aged 95-99 years (3). Between 2000 and 2020, the total number of Chinese people with PAD is expected to increase by 40% from 29.44 million in 2000 to 41.13 million in 2020.

In the early stages, PAD is mostly silent. With the progression of disease, it may manifest as intermittent claudication, pain at rest, non

-healing ulcer and gangrene resulting in lower-extremity amputation [5]. PAD is a major cause of disability, loss of employment, and lifestyle changes, and is a marker for systemic atherosclerotic diseases. Patients with symptomatic PAD have at least a 30% risk of death within 5 years rising to almost 50% within 10 years, resulting primarily from myocardial infarction or stroke [4]. Despite the major health risks associated with PAD, it is generally not recognized by clinicians or the general public in comparison with other cardiovascular diseases. Most individuals with lower extremity PAD are asymptomatic and do not experience recognizable ischemic symptoms until late in the disease progression. However, asymptomatic individuals also have higher risk of adverse cardiovascular events similar to those with symptomatic PAD [6]. Low awareness makes addressing the public health impact of PAD challenging [7]. Many studies have shown that public awareness of PAD is much lower than that of other diseases. It has been reported that awareness of PAD ranged from 20 to 36 %, whereas awareness of other common diseases was more than 60 % in the same population [6-9]. Awareness is important for patients and physicians, and the need for public awareness programs has been highlighted [10, 11]. There is paucity of published literature on public awareness of PAD in Asian countries. It is difficult to reduce the morbidity and mortality of untreated PAD without adequate public awareness of PAD and its risk factors and consequences [7]. Insights into public awareness of PAD will help in developing strategies for behavioral change communication and health promotion. In this study we aimed to assess awareness of PAD among adults in Hong Kong. The survey is designed to measure knowledge of factors that increase the risk for PAD and the clinical risk consequences of having PAD. These data will provide useful information to guide future local public cardiovascular educational efforts.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 or above
* Patients who attend outpatient clinics at the Prince of Wales Hospital

Exclusion Criteria:

* Vulnerable subjects that are illiterate and have severe hearing impairment.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A sample size of 1000 is associated with a margin of error of less than 4.5% and a confidence level of 95%. The study population is weighted by age (into three 20-year categories: 40 to 59, 60 to 79 and ≥80 years of age) and on gender to reflect Hong Kong census estimates for 2016.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Participants' awareness of PAD | 7 months
  Awareness of PAD among adults in Hong Kong will be measured by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No